CLINICAL TRIAL: NCT00204243
Title: Naltrexone Implants Compared to Methadone Maintenance Treatment (MMT) Among Inmates About to be Released From Prison - a Randomized Controlled Trial
Brief Title: Naltrexone Implants vs. MMT Among Inmates in the Norwegian Correctional Services
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Philipp Lobmaier, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Project B: 160115; NCT00520793 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Opiate Addiction
Keywords: naltrexone implant; methadone; inmates; randomized controlled trial
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone; Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone implant (Experimental): Naltrexone implant (GoMedical Inc. 6 months implant)
  Interventions: Drug: Naltrexone
- Methadone (Active Comparator): Methadone Maintenance Treatment
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Naltrexone — surgically implanted naltrexone releasing during 5 to 6 months
  Arms: Naltrexone implant
Drug: Methadone — Methadone maintenance treatment, flexible high dose (80 to 120 mg / Day)
  Arms: Methadone

SUMMARY:
The purpose of this clinical trial is to study the efficacy and safety of naltrexone implants as a relapse prevention for opiate addicted inmates about to be released from prison. The experimental group is compared with a control group that commences methadone maintenance treatment before release.

The hypothesises are that quality of life and criminal behaviour improve significantly in both groups compared to the month before incarceration. The experimental group is going to have significant less days with opioid use compared to the MMT group.

We hypothesize furthermore that the implants can prevent death related to opiate overdose up to 6 months after commenced treatment.

DETAILED DESCRIPTION:
The probability of quick relapse to criminal activity and substance abuse after prison release is high among incarcerated opiate addicts.

We attempt to prevent relapse to opiate abuse by two different means:

Methadone Maintenance Treatment (MMT) versus Naltrexone implants, randomly allocated to two groups by sealed envelopes.

All participants may choose in which group to continue after 6 (and again after 12) months, when the implants supposedly stop releasing naltrexone.

The total treatment period is 18 months, continuation with MMT is optional after study termination.

ELIGIBILITY:
Inclusion Criteria:

* opiate addiction
* living in greater Oslo area

Exclusion Criteria:

* psychosis / major depression, currently not treated
* pregnancy
* liver enzymes: ASAT or ALAT > threefold above upper boundary

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-05; Primary Completion 2008-02 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Drug use: self reported, urin / hair analysis | 6, 12 and 18 months
  Use of heroin and other illicit drugs, self reported and in hair analyses

SECONDARY OUTCOMES:
Distress / depression: BDI and Hopkins SCL-25 | 6, 12 and 18 months
Quality of life, temporary satisfaction with life scale & self report as of ASI | 6, 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Lobmaier, cand. med., Principal Investigator — Unit for Addiction Medicine; Helge Waal, professor, Study Director — Unit for Addiction Medicine, University of Oslo; Michael Abdelnoor, PhD, Study Chair — Ullevål University Hospital, Centre for clinical research; Jørg Mørland, professor, Study Chair — Division of Forensic Toxicology and Drug Abuse; Asbjørg S Christophersen, MD, Study Chair — Division of Forensic Toxicology and Drug Abuse
Locations (1):
- Unit for Addiction Medicine, Oslo, Norway

REFERENCES:
- [Background] Hulse GK, Arnold-Reed DE, O'Neil G, Chan CT, Hansson RC. Achieving long-term continuous blood naltrexone and 6-beta-naltrexol coverage following sequential naltrexone implants. Addict Biol. 2004 Mar;9(1):67-72. doi: 10.1080/13556210410001674112. PMID 15203441
- [Background] Hulse GK, Arnold-Reed DE, O'Neil G, Chan CT, Hansson R, O'Neil P. Blood naltrexone and 6-beta-naltrexol levels following naltrexone implant: comparing two naltrexone implants. Addict Biol. 2004 Mar;9(1):59-65. doi: 10.1080/13556210410001674103. PMID 15203440
- [Background] Hulse GK, Tait RJ, Comer SD, Sullivan MA, Jacobs IG, Arnold-Reed D. Reducing hospital presentations for opioid overdose in patients treated with sustained release naltrexone implants. Drug Alcohol Depend. 2005 Sep 1;79(3):351-7. doi: 10.1016/j.drugalcdep.2005.02.009. PMID 15899557
- [Background] Olsen L, Christophersen AS, Frogopsahl G, Waal H, Morland J. Plasma concentrations during naltrexone implant treatment of opiate-dependent patients. Br J Clin Pharmacol. 2004 Aug;58(2):219-22. doi: 10.1111/j.1365-2125.2004.02122.x. PMID 15255807
- [Background] Bachs L, Waal H. [Naltrexone in the treatment of addiction]. Tidsskr Nor Laegeforen. 2003 Jun 12;123(12):1665-7. Norwegian. PMID 12821984
- [Background] Waal H, Christophersen AS, Frogopsahl G, Olsen LH, Morland J. [Naltrexone implants--a pilot project]. Tidsskr Nor Laegeforen. 2003 Jun 12;123(12):1660-1. Norwegian. PMID 12821982
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Kunoe N, Lobmaier P, Vederhus JK, Hjerkinn B, Gossop M, Hegstad S, Kristensen O, Waal H. Challenges to antagonist blockade during sustained-release naltrexone treatment. Addiction. 2010 Sep;105(9):1633-9. doi: 10.1111/j.1360-0443.2010.03031.x. PMID 20707781